CLINICAL TRIAL: NCT01001013
Title: A Randomized, Open-label, Multiple Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interaction of LC15-0444 and Pioglitazone After Oral Administration in Healthy Male Subjects
Brief Title: Pharmacokinetic Drug Interaction Between LC15-0444 and Pioglitazone After Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: LG Life Sciences, LG Life Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL003
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LC15-0444 200 mg (Experimental): LC15-0444 200 mg
  Interventions: Drug: LC15-0444, Pioglitazone
- Pioglitazone 30 mg (Experimental): Pioglitazone 30 mg
  Interventions: Drug: LC15-0444, Pioglitazone
- LC15-0444 200 mg + pioglitazone 30 mg (Experimental): LC15-0444 200 mg + pioglitazone 30 mg
  Interventions: Drug: LC15-0444, Pioglitazone

INTERVENTIONS:
Drug: LC15-0444, Pioglitazone — LC15-0444 200 mg (100 mg x 2) qd (12 days once daily) Pioglitazone 30 mg (15 mg x 2) qd (12 days once daily) LC15-0444 200 mg (100 mg x 2) qd + pioglitazone 30 mg (15 mg x 2) qd (12 days once daily)

SUMMARY:
The objective of the study is to investigate the drug interaction between LC15-0444 and pioglitazone by comparing the safety, tolerability and pharmacokinetics of LC15-0444 and pioglitazone are administered concomitantly and each alone in healthy male subjects.

DETAILED DESCRIPTION:
This study is a randomized, open-label, three-treatment, three-period, three-sequence and crossover design in healthy volunteers to evaluate tolerability, safety and pharmacokinetics after the multiple administration of LC15-0444 and pioglitazone concomitantly or each alone.

Eligibility for participation of this study will be determined by demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 3 weeks(-21 d ~ -2 d) before drug administration(1 d). Eligible subjects will be randomized to one of three sequence groups.

According to the characteristics of anti-diabetic drugs, it is expected to be administered with other anti-diabetic drugs. Therefore, Drug-Drug Interaction with Pioglitazone should be identified in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 20 and 45 years at screening
2. Subjects with Body Mass Index (BMI) between 18.0(inclusive) and 27.0 kg/m2 (exclusive); and a total body weight between 55 kg (inclusive) and 90 kg (exclusive). BMI(kg/m2) = body weight(kg)/{height(m)}2.
3. Subjects with fasting plasma glucose (FPG) level of 70-125 mg/dL (both inclusive) at the time of screening.
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.

Exclusion Criteria:

1. Subjects with evidence or history of clinically significant hepatic (including carrier of viral hepatitis), renal, neurologic (mood disorder, obsessive-compulsive disorder etc.), immunologic, pulmonary, endocrine, hematological, neoplastic, cardiovascular or psychiatric disease.
2. Subjects with evidence or history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis etc.) or surgery (except appendectomy and herniotomy) possibly affecting drug absorption.
3. Subjects with history of hypersensitivities including drug allergies (caused by aspirin, antibiotics, etc.), or history of clinically significant hypersensitivities.
4. Subjects who meet the following criteria at the time of the screening examination; Serum AST(SGOT) or ALT(SGPT): > 1.5 times upper normal limit Creatinine clearance calculated by Cockcroft-Gault equation

   * < 80 mL/min Clinical significant abnormalities on ECG including 12-lead ECG demonstrating QTc >450 msec at screening or any rhythms except for sinus rhythm
5. Subjects who show the following vital sign results at sitting position after resting for 3 min; SBP: ≤ 100 mmHg or ≥ 150 mmHg DBP: ≤ 60 mmHg or ≥ 95 mmHg
6. Subjects with history of drug abuse or a positive urine result in drug screen for drug abuse or cotinine.
7. Subjects who have taken any prescribed medicines or herbal medicines within 2 weeks before the first administration of the investigational product, any non-prescribed medicines or vitamin supplements within 1 week before the first administration of the investigational product. (If other conditions are satisfied, subjects may be eligible for the trial by the investigator's judgment.)
8. Subjects who have participated in any other clinical trial within 2 months before the first administration of the investigational product.
9. Subjects who have donated a unit of blood within 2 months or blood components within 1 month before the first administration of the investigational product.
10. Subjects who consume more than 21 units of alcohol per week (1 unit = 10 g of pure alcohol) or unable to abstain from drinking throughout the trial.
11. Smokers (except for those who quit smoking for at least 3 months the first administration of the investigational product)
12. Subjects who take caffeine-containing or grapefruit-containing products within 3 days before the first administration of the investigational product.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss, Cmax,ss of LC15-0444 and pioglitazone | During all dosing visits

SECONDARY OUTCOMES:
Tmax,ss, t1/2, CL/F, Aeτ,ss, CLR, Ctrough,ss of LC15-0444 and pioglitazone AUCτ,ss, Cmax,ss, metabolic ratio of LC15-0444, Pioglitazone metabolites AUC,ss, Cmax,ss, metabolic ratio of pioglitazone metabolites | During all dosing visits

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim SE, Yi S, Shin KH, Kim TE, Kim MJ, Kim YH, Yoon SH, Cho JY, Shin SG, Jang IJ, Yu KS. Evaluation of the pharmacokinetic interaction between the dipeptidyl peptidase IV inhibitor LC15-0444 and pioglitazone in healthy volunteers. Int J Clin Pharmacol Ther. 2012 Jan;50(1):17-23. doi: 10.5414/cp201568. PMID 22192641